CLINICAL TRIAL: NCT01591798
Title: Clinical Assessment of Laparoscopic and Robotic Surgery for Rectal Cancer - Randomized Phase II Trial
Brief Title: Efficacy Study of Robotic Surgery for Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji Won Park, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-CTS603
Record Dates: First submitted 2012-03-16; First posted 2012-05-04 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Rectal Neoplasm
Keywords: Rectal cancer; Robotic surgery; Laparoscopic surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

ARMS (2):
- Robotic surgery (Experimental): Proctectomy using robot
  Interventions: Procedure: Robotic surgery
- Laparoscopic surgery (Active Comparator): Conventional laparoscopic rectal resection
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Robotic surgery — Robotic assisted rectal resection
  Other Names: da Vinci Surgical System
  Arms: Robotic surgery
Procedure: Laparoscopic surgery — Laparoscopic assisted rectal resection
  Arms: Laparoscopic surgery

SUMMARY:
After introducing minimally invasive surgery, robotic surgery has been increasingly used in colorectal cancer. However, there is a few prospective study for robotic surgery. The aim of this trial is to evaluate the effectiveness and safety of robotic surgery in mid or low rectal cancer.

DETAILED DESCRIPTION:
This study was designed as randomized phase II trial (laparoscopic versus robotic). The primary end point is quality of mesorectal excision.

ELIGIBILITY:
Inclusion Criteria:

* mid or low rectal cancer (within 9cm from anal verge)
* pathologically proven as adenocarcinoma
* written informed consent
* no severe functional disability in lung and heart

Exclusion Criteria:

* invading adjacent organ
* distant metastasis (lung, liver, brain, bone, distant lymph nodes etc.)
* lateral pelvic lymph node metastasis
* Have severe concomitant disease that might limit compliance or completion of the protocol.
* Have any other malignancy that might impact 5-year survival or might be potentially confused with rectal cancer.
* If female, be pregnant or breast feeding.
* Hereditary colorectal cancer (HNPCC, FAP etc)
* emergency operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of mesorectal excision | 7days after surgery (Pathologic report)
  Evaluating the quality of mesorectal excision in rectal specimen according to the criteria suggested by Nagtegaal ID, et al. (J Clin Oncol. 2002;20:1729-34)

SECONDARY OUTCOMES:
Short-term postoperative outcome | Within postoperative 30 days
Sexual and urinary function, Quality of life, Anorectal function | Baseline, postop 3 weeks, 3months, 12 months, 24 months, 36 months
  IIEF, FSFI, IPSS, EORTC C30, CR38, FISI, MSKCC bowel fuction tool, Manometry
Long-term outcome | Postoperative 36 months
  3 year disese-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Park, Dr., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea